CLINICAL TRIAL: NCT05097976
Title: An Oral Methylprednisolone Taper Within a Multimodal Analgesic Regimen After Total Knee Arthroplasty: a Double-Blind Randomized Placebo-Controlled Trial
Brief Title: Medrol Dosepak for Outpatient Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Professor of Orthopedic Surgery, Chief Division of Adult Reconstruction, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21090203
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Methylprednisolone; acute postoperative pain; acute function; opioid consumption; complications following total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigator (surgeon) and participant (patient) will be blinded to whether they are discharged with a placebo or treatment (oral corticosteroid).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylprednisolone taper (Experimental): Methylprednisolone taper - 21 x 4mg tablets beginning on POD 1
  Interventions: Drug: Methylprednisolone
- Placebo taper (Placebo Comparator): 2.Placebo taper - 21 sugar tablets beginning on POD 1 with standard management
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — 21 x 4mg tablets beginning on POD 1
  Other Names: medrol dosepak
  Arms: Methylprednisolone taper
Drug: Placebo — 21 sugar tablets beginning on POD 1 with standard management
  Arms: Placebo taper

SUMMARY:
The purpose of this study is to evaluate the efficacy of an oral methylprednisolone taper on acute postoperative pain, function, opioid consumption, nausea, and complications following outpatient total knee arthroplasty (TKA). We hypothesize that administration of an oral methylprednisolone taper starting on postoperative day 1 (POD 1) following TKA will be associated with improved pain and decreased opioid use, nausea, and complications at POD1-7, as compared to similar patients who receive placebo. Additionally, those taking methylprednisolone will report decreased pain and greater objective functional outcomes at 3 and 6 weeks postoperatively as compared to controls.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) has been associated with severe pain in the acute postoperative period. Studies have demonstrated highest pain scores on POD 1 following TKA, however over 50% of patients describe the first two weeks at home as the most painful period of recovery marked by moderate to severe pain. This is an important finding as higher levels of acute pain have been associated with chronic opioid use, disturbed sleep, and impaired early mobilization, which can prolong recovery time and increase rates of adverse events, including venous thromboembolism.

Therefore, extensive research in pain management has been conducted with the purpose of reducing acute postoperative pain. This is of particular interest because over the past two decades average length of hospital stay has decreased while rates of outpatient TKAs with same day discharge has increased. A multimodal pain regimen enables the on-boarding of several medications, including anesthesia and analgesics working at varied pathways to target pain and inflammation, and has proven to be efficacious. This not only decreases patient reported pain scores but is also associated with improved sleep and functional recovery. Despite efficacious multimodal pain regimens, including periarticular injection cocktails, rebound pain in the early postoperative period and medication-induced nausea and vomiting can be problematic.

Corticosteroids are potent anti-inflammatory and pain pathway modulators, and therefore have become an important component of multimodal pain regimens. Corticosteroids have been shown to decrease postoperative levels of inflammatory mediators, such as IL-6 and C-reactive protein. Corticosteroids also block the synthesis of prostaglandins, a nociceptive pain receptor sensitizer and inflammatory mediator that is associated with edema via increased vascular permeability.

The administration of perioperative steroids to mitigate potential impairments in postoperative TKA recovery has been studied extensively in the orthopedic literature. The addition of corticosteroids to multimodal pain regiments, including systemic corticosteroids or perioperative periarticular joint cocktails, has demonstrated improved acute postoperative pain scores function and decreased opioid use without an increase in adverse outcomes, as compared to controls.

Researchers have investigated the effect of additional doses of corticosteroids in the immediate postoperative period. Administration of IV dexamethasone 24 hours postoperatively correlated with lower acute opioid and antiemetic use, and improved pain scores, nausea, length of stay and range of motion, as compared to controls or perioperative corticosteroids alone. The addition of a second postoperative corticosteroid dose, at 24 and 48 hours, have been associated with even greater improvements in pain and function scores, without an increase in complications.

The addition of a methylprednisolone taper within a standard multimodal pain regimen in the immediate postoperative period has been evaluated in other orthopedic subspecialties. A methylprednisolone taper following lumbar laminectomy and distal radius repair demonstrated acute reductions in patient reported pain scores, without an increase in adverse events. The current literature supports these findings, demonstrating the safety of short term and low dose corticosteroid treatments, including a methylprednisolone taper.

To the best of our knowledge, no prior study has compared the administration of a methylprednisolone taper to a placebo in the immediate postoperative period following TKA. Therefore, the purpose of this double-blind randomized placebo-controlled trial is to evaluate the efficacy of a methylprednisolone taper within a standard postoperative multimodal pain regimen. The authors predict improved pain and decreased opioid use and nausea from POD 1 to POD 7, as well as improved pain, function, and complication rate at 3- and 6-weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing primary TKA with a diagnosis of osteoarthritis

  •≥ 18 years old
* Willingness to undergo randomization

Exclusion Criteria:

* Reported chronic corticosteroid or opiate use
* Suspected or confirmed periprosthetic joint infection
* Revision TKA
* Primary diagnosis other than osteoarthritis, including avascular necrosis, fracture, or post-traumatic arthritis
* American Society of Anesthesiologists (ASA) score ≥ 4
* Reported history of liver disease, renal disease, or diabetes mellitus
* Current systemic fungal infection or other local infection
* Immunocompromised or immunosuppressed
* Current peptic ulcer disease
* History of hypothyroidism, psychosis, heart failure, myasthenia gravis, ocular herpes simplex virus, or systemic sclerosis
* Women with reported current pregnancy
* Known hypersensitivity to methylprednisolone

  •≤ 18 years old
* Inability to take oral medications
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption at one-week postoperative | one week
  Relative difference in cumulative opioid consumption at Post-op day 7, measured in morphine equivalents.

SECONDARY OUTCOMES:
Patient reported outcome measures: Daily Visual Analogue Scale for Pain | Week 1
  Using Daily Visual Analogue Scale (VAS) pain score, scale of 1 to 10, 10 being the worst
Patient reported outcome measures : Daily Visual Analogue Scale for Pain | 3 weeks
  Using Daily Visual Analogue Scale (VAS) pain score, scale of 1 to 10, 10 being the worst
Patient reported outcome measures: Daily Visual Analogue Scale for Pain | 6 weeks
  Using Daily Visual Analogue Scale (VAS) pain score, scale of 1 to 10, 10 being the worst
Patient reported outcome measures: Daily Visual Analogue Scale of nausea | Postoperative days 1 through 7 (week one)
  Daily visual analogue scale- nausea score, scale of 1 to 10, 10 being the worst
Patient reported outcome measures: vomiting episodes | Postoperative days 1 through 7 (week 1)
  Number of vomiting episodes, patient reported
Patient reported outcome measures: hours of sleep | Postoperative days 1 through 7 (week one)
  Number of hours slept- patient reported
Clinical outcome: range of motion | Preoperatively
  range of motion of knee
Clinical outcome: range of motion | 3 weeks after treatment
  range of motion of knee
Clinical outcome: range of motion | 6 weeks after treatment
  range of motion of knee
Patient reported outcome measures: knee society score | Preoperatively
  Knee society score (KSS) survey
Patient reported outcome measures: knee society score | 3 weeks after treatment
  Knee society score (KSS) survey
Patient reported outcome measures: knee society score | 6 weeks after treatment
  Knee society score (KSS) survey

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush Oak Brook Outpatient Center, Oak Brook, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided